CLINICAL TRIAL: NCT01918891
Title: Center for Stroke Disparities Solution (CSDS) Project II: Community Transitions Intervention (CTI)
Brief Title: Center for Stroke Disparities Solution - Community Transitions Intervention
Acronym: CSDS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Visiting Nurse Service of New York (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); NYU Langone Health (Other); Hebrew Home at Riverdale (Other); Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: I12-004; 1U54NS081765 (NIH)
Record Dates: First submitted 2013-08-05; First posted 2013-08-08 (Estimated); Last update posted 2019-10-01 (Actual); Status verified 2019-09

CONDITIONS: Hypertension; Stroke; Transient Ischemic Attack
Keywords: stroke; transient ischemic attack; High blood pressure; Hypertension
MeSH Terms: conditions — Hypertension; Stroke; Ischemic Attack, Transient | interventions — Nurse Practitioners

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Usual Home Care (No Intervention): Regardless of study arm, all patients will receive usual home health services: a physician-ordered plan of care; skilled nursing and/or therapy services as prescribed by the MD; patient education, monitoring and hands-on care; and home health aide services depending on functional deficits and availability of unpaid caregivers.
- Nurse Practitioner + Health Coach (Experimental): The NP + HC arm will include the same protocol as the NP only arm plus 30 additional days of support. The HC will pick up the case after the initial 30 days and follow up with the plan of care jointly established by the patient, NP and HC. The focus will be on ongoing self-management coaching, providing preparation support for physician visits, and linking patient to additional community resources, as needed.
  Interventions: Behavioral: Nurse Practitioner Only; Behavioral: Nurse Practitioner + Health Coach
- Nurse Practitioner Only (Experimental): The NP only program will provide a 30 day intervention via in-home and telephone encounters for patients randomized to this group. In the first 30 days post-enrollment the NP will focus on medical case management and coordination with primary care providers and specialists, provide self-management coaching, and intervene if gaps in care are identified - all with a focus on BP reduction and preparing the patient for ongoing BP maintenance.
  Interventions: Behavioral: Nurse Practitioner Only

INTERVENTIONS:
Behavioral: Nurse Practitioner Only
  Arms: Nurse Practitioner + Health Coach; Nurse Practitioner Only
Behavioral: Nurse Practitioner + Health Coach
  Arms: Nurse Practitioner + Health Coach

SUMMARY:
The Stroke CTI study is a 3 arm randomized, controlled trial designed to assess the effectiveness of a nurse practitioner (NP) only and a NP and health coach (HC) community transitions intervention (CTI) in reducing secondary stroke risk by helping patients lower their systolic blood pressure.

DETAILED DESCRIPTION:
Targeted study participants are Black and Hispanic patients with a history of stroke and a current systolic blood pressure (BP) above JNC7 recommended range (>=140 mmHg) who recently entered home care service. The NP only program will provide a 30 day intervention while the NP/HC team will provide 3 months of support via in-home and telephone encounters for patients randomized to one of these groups. In the first 30 days post-enrollment the NP will focus on medical case management and coordination with primary care providers and specialists, provide self-management coaching, and intervene if gaps in care are identified - all with a focus on BP reduction and preparing the patient for ongoing BP maintenance. As applicable, the HC will pick up the case after 30 days and follow up with the plan of care jointly established by the patient, NP and HC. The focus will be on ongoing self-management coaching, providing preparation support for physician visits, and linking patient to additional community resources, as needed.

ELIGIBILITY:
Inclusion Criteria:

* Newly admitted to the VNSNY post acute care program
* 21 years of age or older
* Black and/or Hispanic
* Speaks English or Spanish
* History of stroke or transient ischemic attack (TIA)
* Hypertension diagnosis
* Average screening systolic BP >= 140 mmHg
* Is available to participate in intervention activities during the study timeframe if randomized to treatment group

Exclusion Criteria:

* Dialysis
* End stage renal disease
* Kidney transplant
* Severe heart failure
* Significant cognitive impairment. Unable to provide informed consent, accurate self-report, and/or unable to participate effectively in intervention
* Significant verbal speech impairment. Unable to participate in intervention telephone sessions
* Patients with upper arm circumference outside of valid use parameters for the automated device used for eligibility screening

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 495 (Actual)
Dates: Start 2012-09 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Reduction of systolic blood pressure | Baseline to 3 and 12 months.
  Patients randomized to the NP only and the NP+HC transitional care interventions will have greater 3 and 12 month reduction in SBP than patients in Usual Home Care.

SECONDARY OUTCOMES:
Cost-effectiveness of NP-only and NP+HC relative to UHC | VNSNY home care admission to 3 and 12 months post admission
  Both interventions will be more costly but more cost-effective than usual home care.
Influence on post-stroke patients' function and health-related quality of life (QoL) | Baseline to 3 and 12 months
  Both interventions will yield significant comparative improvements in function and health-related QoL; NP+HC will be more effective than NP-only.

OTHER OUTCOMES:
Moderators and mediators that may affect treatment outcomes | Baseline to 3 and 12 months
  Exploratory aim to examine potential moderating/mediating variables which may include: moderators - race/ethnicity (i.e., Black/Hispanic differences), baseline HTN severity (Stage I vs. Stage II); mediators - 1) changes in health behaviors (i.e., diet, physical activity, weight loss, medication adherence); and 2) antihypertensive medication intensification (i.e., adding, changing dose, or changing class of medications).

CONTACTS AND LOCATIONS:
Overall Officials: Penny H Feldman, PhD, Principal Investigator — Visiting Nurse Service of New York
Locations (1):
- Visiting Nurse Service of New York, New York, New York, United States

REFERENCES:
- [Derived] Osakwe ZT, Barron Y, McDonald MV, Feldman PH. Effect of Nurse Practitioner Interventions on Hospitalizations in the Community Transitions Intervention Trial. Nurs Res. 2021 Jul-Aug 01;70(4):266-272. doi: 10.1097/NNR.0000000000000508. PMID 34160182
- [Derived] Feldman PH, McDonald MV, Trachtenberg M, Trifilio M, Onorato N, Sridharan S, Silver S, Eimicke J, Teresi J. Reducing Hypertension in a Poststroke Black and Hispanic Home Care Population: Results of a Pragmatic Randomized Controlled Trial. Am J Hypertens. 2020 Apr 1;33(4):362-370. doi: 10.1093/ajh/hpz148. PMID 31541606
- [Derived] Feldman PH, McDonald MV, Trachtenberg MA, Schoenthaler A, Coyne N, Teresi J. Center for stroke disparities solutions community- based care transition interventions: study protocol of a randomized controlled trial. Trials. 2015 Jan 27;16:32. doi: 10.1186/s13063-015-0550-3. PMID 25622823
- See also: NYU School of Medicine - Center for Stroke Disparities Solutions — http://pophealth.med.nyu.edu/divisions/chbc/research/csds